CLINICAL TRIAL: NCT04327895
Title: Surgery in Context of Terrorist Attack : Report of the 121st Annual Congress of French Association of Surgery
Brief Title: Surgery in Context of Terrorist Attack : a Survey of French Surgeons
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Association Francaise de Chirurgie (Other)
Responsible Party: Sponsor
Other Study IDs: AFC
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2019-03

CONDITIONS: Trauma Injury; War Injury; Surgical Procedure, Unspecified
Keywords: need for surgical training; surgery and terrorist attack
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: evaluation of the need for training — analyse of results of survey

SUMMARY:
The aim of the study is to assess the surgical knowledge of French Surgeons in cas of Terrorist Attack.

DETAILED DESCRIPTION:
Survey was sent by email to French Surgeons affiliated to French Association of General Surgeons.

First series of questions are relative to age, qualification, usual surgical practice, in order to define different "surgical profiles".

Second series of questions are relative to knowledge in the field of knowledge about trauma and massive casualties surgery.

Third series of questions are relative to the feeling of easiness in case of various situations involving severe trauma and massive casualties.

Results are analyzed in order to assess the need for learning and training in the field of trauma and massive casualties surgery.

ELIGIBILITY:
Inclusion Criteria:

* French Licensed and Resident Surgeons

Exclusion Criteria:

* Medical Doctor, not Resident

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French General Surgeons who are working as Resident or Licensed Surgeons in Public or Private Hospitals, and who are amenable to manage massive casualties due to Terrorist Attack
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
assessing the knowledge and the skills of general surgeons in the field of trauma surgery | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Balandraud, MD, Study Director — Direction Centrale du Service de Santé des Armées
Locations (1):
- Military Hospital, Toulon, France

IPD SHARING:
Plan to Share IPD: No
No sharing plan